CLINICAL TRIAL: NCT00115128
Title: Open-Label Trial of Peripheral Blood Progenitor Cell (PBPC) Mobilization by Filgrastim in Normal Donors
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20020143; NCT00108966 (obsolete NCT alias)
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Normal PBPC Donors
Keywords: normal PBPC donors
MeSH Terms: interventions — Filgrastim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — none collected

GROUPS / COHORTS (1):
- Filgrastim: Normal donors being treated with filgrastim for PBPC mobilization and collection
  Interventions: Drug: filgrastim

INTERVENTIONS:
Drug: filgrastim — Normal donors being treated with filgrastim for PBPC mobilization and collection

SUMMARY:
The purpose of this study is to clinically evaluate the spleen during PBPC mobilization by filgrastim in normal donors.

ELIGIBILITY:
Inclusion Criteria: - Eligible to be PBPC donor for allogeneic transplantation as determined by local institution Exclusion Criteria: - History of splenectomy - Previous PBPC mobilization attempts - Previous treatment with GCSF or GMCSF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Normal donors
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2003-11; Primary Completion 2007-05 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Spleen fold change measured by ultrasound | Before, during, and through 1 week post-PBPC mobilization and collection

SECONDARY OUTCOMES:
Spleen change associations with filgrastim dose and hematologic variables | Before, during, and through 1 week post-PBPC mobilization and collection

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Stiff PJ, Bensinger W, Abidi MH, Gingrich R, Artz AS, Nademanee A, Hansen KS, Sobczak C, Cutler C, Bolwell B, Shore TB, Lazarus HM, Yeager AM, Lovelace W, Guo M, Dreiling L. Clinical and ultrasonic evaluation of spleen size during peripheral blood progenitor cell mobilization by filgrastim: results of an open-label trial in normal donors. Biol Blood Marrow Transplant. 2009 Jul;15(7):827-34. doi: 10.1016/j.bbmt.2009.03.015. PMID 19539214
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_06_G-CSF_20020143.pdf